CLINICAL TRIAL: NCT05100563
Title: Participant(s) With Autism and High Pain Tolerance Treated With High Dose Naltrexone
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: aUTISM01
Record Dates: First submitted 2020-10-22; First posted 2021-10-29 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Naltrexone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 50 mg naltrexone — Medication combined with twice a week psychotherapy

SUMMARY:
High dose naltrexone with response gauged by pain tolerance as measured by the cold pressor test may help treat autism.

DETAILED DESCRIPTION:
Clinical Trial: Cause and Treatment of High Opioid Tone Autism Key Words: autism, neurobiological systems engineering, opioid tone, cold pressor time, clinical trial Abstract Introduction: Neurobiological systems engineering models are useful for treating patients. We show a model of "high opioid tone" autism and present a hypothesis about how autism is caused by administration of opioids during childbirth.

Main Symptoms: Clinical diagnosis of autism in a 25 year old man was confirmed by a Social Responsiveness Scale (SRS) self - rating of 79, severe, and a Social Communications Questionnaire (SCQ - 2) by the patient's father scoring 27. Cold pressor time is a measure of pain tolerance obtained by having the subject submerge their normal forearm in a painful ice water bath. Cold pressor time (CPT) was 190 seconds - unusually long, consonant with the high pain tolerance of autism.

Therapeutic Intervention and Outcome Measure:

Primary Outcome Measure is the Cold Pressor Time (CPT). At naltrexone 50 mg/day CPT fell to 28, repeat 39 seconds.

Secondary outcome measures are Social Responsiveness Scale (SRS) and Social Communications Questionnaire (SCQ-2). SRS fell to 54 and SCQ - 2 to 9; both non - significant for autism.

Change in relatedness was experienced ambivalently, understood as feelings never before experienced - causing pain. Non - compliance with naltrexone was followed by cutting open his palm and drinking alcoholically. Transference focused psychotherapy has helped him remain naltrexone - compliant while he works on issues of identity and relatedness.

Conclusion: The model suggests studies that could be conducted to both prevent and treat this form of autism.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of autism -

Exclusion Criteria: Lack of ability to give informed consent

-

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adults with autism spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
improvement of social responsiveness scale (SRS) and social communication questionnaire (SCQ) | After two weeks at optimal naltrexone dose
  evaluation by patient at baseline and follow up of SRS and his father SCQ

SECONDARY OUTCOMES:
Cold Pressor Time | After a week on optimized naltrexone dose with repeat two weeks later
  At baseline and after optimized naltrexone dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No